CLINICAL TRIAL: NCT01218568
Title: Rifaximin Plus Lactulose Versus Lactulose Alone for the Treatment of Hepatic Encephalopathy: a Double Blind Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS HE-01
Record Dates: First submitted 2010-10-05; First posted 2010-10-11 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-06

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin; Lactulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifaximin plus lactulose (Experimental)
  Interventions: Drug: Rifaximin plus lactulose
- lactulose (Active Comparator): 30-60ml/day
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Rifaximin plus lactulose — Rifaximin 400 mg three times a day Lactulose 30-60 ml in two or three divided doses.
  Arms: Rifaximin plus lactulose
Drug: Lactulose — Lactulose 30-60 ml in two or three divided doses.
  Arms: lactulose

SUMMARY:
The study will be double blind with respect to rifaximin, and randomization will be performed using tables of computer-generated random numbers. All subjects will be followed up till the recovery of HE (primary end point) or 10 days whichever is earlier. In the Lactulose group (group A) patients will receive 30-60 ml of lactulose in 2 or 3 divided doses so that patient passes 2-3 semisoft stools per day along with placebo . In the lactulose plus rifaximin group (group B) patients will receive cap rifaximin 400mg three times a day along with lactulose. Primary endpoints will be recovery of overt HE patients who will not recover from HE after 10 days will be continued on the same treatment. Total duration of the study is 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Age 18-80
* Hepatic encephalopathy grade II-IV
* Informed consent

Exclusion Criteria:

1. Degenerative CNS disease or major psychiatric illness
2. Serum creatinine > 1.5 mg/dl
3. Active alcohol intake <4 weeks prior to present episode
4. Others metabolic encephalopathies
5. Hepatocellular Carcinoma
6. Severe comorbidity such as CHF, Pulmonary disease, Neurological & Psychiatric problems impairing quality of life

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Reversal of hepatic encephalopathy | 10 days

SECONDARY OUTCOMES:
Death | 10 days
duration of hospital stay | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India